CLINICAL TRIAL: NCT04545203
Title: Effects of Slow-Stroke Back Massage on Chemotherapy-releated Fatigue in Breast Cancer Patients: An Assessor-blinded, Parallel Group, Randomized Controlled Trial
Brief Title: Effects of Slow-Stroke Back Massage on CRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Pinar Zorba Bahceli, PhD RN, Asistant Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017/62
Record Dates: First submitted 2020-09-05; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Chemotherapy-releated Fatigue
Keywords: Chemotherapy-releated fatigue; Slow-stroke back massage; Nursing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow-Stroke Back Massage Group (Experimental)
  Interventions: Other: Slow-stroke back massage
- Control group (No Intervention)

INTERVENTIONS:
Other: Slow-stroke back massage — Slow-stroke back massage was performed to the breast cancer patients in intervention group. The SSBM sessions were administered 10 minutes before and after chemotherapy treatment.The SSBM was applied for 20 minutes in total, on each cycle. The intervention group received 20-minute SSBM sessions 3 chemotherapy cycle in addition to the routine care.
  Arms: Slow-Stroke Back Massage Group

SUMMARY:
Chemotherapy-related fatigue (CRF) is common in patients with breast cancer and it can be seen between 27% and 96% depending on the stage of cancer and treatment method. At the same time, CRF is reported as the most important symptom that reduces the functional capacity of patients with breast cancer and impairs their quality of life. For this reason, there is a need for an intervention that could decrease or prevent of CRF in breast cancer patients. In the literature, it is stated in the evidence-based guidelines that massage, which is one of the non-pharmacological methods, can be effective in CRF management.

DETAILED DESCRIPTION:
This an assessor-blinded,parallel group randomized controlled trial aimed that investigating the effect of slow-stroke back massage on CRF in breast cancer patients.This trial was conducted in the chemotherapy outpatient clinic of University Hospital located in Turkey. All patients were women who received Adriamycin-Cyclophosphamide (AC)/ Cyclophosphamide-Adriamycin-5 Fluoro-uracil (CAF) regimens every 21 days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older women,
* Stages II or III breast cancer patients who had received at least 1 cycle of chemotherapy and were scheduled to receive 3 more cycles,
* Receiving one of the adriamycin-cyclophosphamide/cyclophosphamide-adriamycin-5-fluorouracil (AC/CAF) chemotherapy protocols,

Exclusion Criteria:

* With metastasis
* Having open wounds and edema on the upper limbs and back
* Using any complementary and alternative (CAM) treatment method to prevent fatigue during administration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Brief Fatigue Inventory | It was filled before and after the 2nd, 3rd and 4th chemotherapy cycles (each cycle is 21 days). Changes in the Brief Fatigue Inventory scores were recorded before and after each three cycles.
  The Brief Fatigue Inventory consisting of 10 items. First item evaluates whether patients with cancer experienced fatigue differently than usual in the previous week. Inventory includes items assessing general fatigue levels of patients (fatigue felt at the time of the interview, fatigue in general and the worst fatigue suffered in the past 24 hours) and the interference of fatigue with daily activities (general activity, mood, walking ability, work life, relationships with other people, the joy of life) in the past 24 hours. Scoring ranges between "0" and "10", "0" indicating no impact at all and "10" indicating the highest level of impact. Global Brief Fatigue Inventory score is calculated by taking the arithmetic mean of other 9 items. The total score to be obtained from the inventory is between 0 and 90. Çınar et al. performed the validity and reliability study of the Turkish version of Brief Fatigue Inventory and the internal consistency of the scale was determined to be 0.98.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Bakircay University Health Sciences Faculty, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No